CLINICAL TRIAL: NCT02965690
Title: Comparison of in Vivo Kinematics of Different Implants in ACL-sacrificing vs. Medially Stabilized Arthroplasty (Implant Design Study)
Brief Title: Kinematics of Contemporary Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse More and Romsdal Trust (Unknown)
Responsible Party: Principal Investigator, Stephan M Rohrl, PhD, MD, orthopaedic consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 424444-2
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty (TKA); Total knee replacement (TKR); Knee kinematics; Dynamic RSA; Fluoroscopy; Fluoroscopic Roentgen Stereophotogrammetric Analysis (FRSA); Medial pivot; Medially stabilized
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-group, non-blind, randomized clinical study
Masking Description: Non-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zimmer Biomet NexGen CR (Active Comparator): Patients receive a Zimmer Biomet NexGen Total Knee Replacement
  Interventions: Procedure: Zimmer Biomet NexGen CR
- Medacta International GMK Sphere (Active Comparator): Patients receive a Medacta International, GMK Sphere Total Knee Replacement
  Interventions: Procedure: Medacta International GMK Sphere

INTERVENTIONS:
Procedure: Zimmer Biomet NexGen CR — Total Knee Replacement
  Arms: Zimmer Biomet NexGen CR
Procedure: Medacta International GMK Sphere — Total Knee Replacement
  Arms: Medacta International GMK Sphere

SUMMARY:
Total joint replacement is an efficacious treatment for osteoarthritis of hips and knees. Both total knee replacement (TKR) and total hip replacements (THR) have excellent implant survivorship. However, patient satisfaction is lower in TKR than THR. A possible cause of the discrepancy is the unnatural knee kinematics after TKR. Various implant designs have been developed to solve the problem. However, most of the designs are based on experimental data and not on in vivo kinematics. In this study, we will analyze the in vivo kinematics of the Global Medacta Knee Sphere (GMK Sphere) implant and compare it with a well documented design and implant (NexGen Cruciate Retaining (CR), Zimmer Biomet). We assume our study will contribute to the development of more satisfying knee implants.

DETAILED DESCRIPTION:
Worldwide the number of patients requiring treatment for osteoarthritis is increasing due to increasing obesity, an ageing population and a high demanding younger population. Learmonth describes hip arthroplasty as the "operation of the century" because patients are highly satisfied with pain relief and function after the procedure. Knee arthroplasties have in recent years also shown promising results and have surpassed hip arthroplasty in frequency in western countries. However, patient satisfaction is not as high. Reported problems are insufficient function and persistent pain. On the other hand, knee arthroplasties are increasingly implanted in younger and more active patients who require high function and quality of life. Improvement of results after knee arthroplasty is therefore an urgent issue in the field of orthopaedic research.

Knee kinematics and implant designs:

A possible cause of lower function of replaced knees is the unnatural postoperative knee kinematics. The kinematics of replaced knees are closely related to their function. Studies show that replaced knees with excellent flexion angles have kinematic similarities to normal knees and malalignments of implants can cause postoperative pain.

Compared to the hip joint which is a simple ball-and-socket joint, the kinematics of knee is more complex. Native knee kinematics are a combination of a rolling and gliding motion of the femoral condyles and rotation of the tibia, where roll back of the lateral femoral condyle is larger than medially. Roll back is important for high degrees of flexion. Native knee kinematics are not fully understood, but the anterior cruciate ligament (ACL) seems to be an integral part, as knees without a functioning ACL show decreased roll back. Based on the kinematics of the normal knee joint, various attempts have been made on the design of knee implants to reconstruct normal kinematics after replacement surgery, but in knee osteoarthritis the ACL and posterior cruciate ligament (PCL) is often deficient as they are damaged by inflammation. Therefore, there are three concepts regarding the retaining of these ligaments in knee replacement surgery. 1: Sacrifice both the ACL and PCL, 2: Retain the PCL (cruciate retaining (CR) design), 3: Retain both the ACL and PCL (bicruciate-reataining design).

The function of the cruciate ligaments can be mimicked by different designs of the tibial insert. The CR design has been widely used in the northern countries, especially the Zimmer Biometri NexGen CR implant in Norway. There are migration data for the NexGen implant with high precision measurements available in the literature. However, the NexGen CR implant does not retain the ACL and does not mimic natural knee kinematics.

The tibial insert of the medially stabilized implant design (Medacta International, GMK Sphere) has a constrained medial "ball in socket" joint and at the same time allows lateral anterioposterior movement (roll back). This new design was developed by a group of dedicated researchers. The design intention is to resemble the native kinematics of the knee by mimicing the function of the cruciate ligaments and at the same time allow for lateral anterioposterior movement (rollback). Theoretically, knee implant designs, which retain the function of cruciate ligaments are predicted to have the closest kinematics to normal knees compared to other designs and to have the potential to achieve the highest patient satisfaction.

Analytical Method:

Radiostereometric Analysis (RSA) has been used in orthopedic research fields since 1970s. The original application of this method was for the evaluation of implant migration (i.e. fixation) and polyethylene wear of artificial joints using static X-ray pictures. When combining RSA with fluoroscopy, we get Fluoroscopic Roentgen Stereophotogrammetric Analysis (FRSA), a method with high accuracy and precision. Few implants have been analysed kinematically in vivo. We plan to investigate the knees during in vivo motion and weight-bearing using FRSA.

Purpose of the study:

The aim of this study is to analyse the in vivo kinematics of a medially stabilized knee arthroplasty implant (GMK Sphere) and to compare it with a well known design (Nexgen CR, Zimmer Biomet) by using FRSA.

By using flat panel fluoroscopy, we will document and compare the kinematics of the two implants in all 6 degrees of freedom (DOF).

26 patients will be randomized into two groups, one will receive the NexGen CR prosthesis, the other group the GMK Sphere.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with knee osteoarthritis

Exclusion Criteria:

1. Preoperative severe deformity (Femoro-tibial angle < 175°or > 190° measured on a full-length leg image at weight bearing)
2. Preoperative flexion contracture more than 15°
3. Preoperative limited range of motion under anesthetics (less than 110°)
4. Less than 50 or more than 75 years of age at the time of surgery
5. Use of walking aids because of other musculoskeletal and neuromuscular problems
6. Preoperative diagnosis other than osteoarthritis and avascular necrosis (e.g. rheumatoid arthritis, tumors)
7. Revision arthroplasty
8. Obesity with BMI>35
9. Impaired collateral ligaments
10. Postoperative KOOS score less than 80
11. Malposition of femoral and tibial implants (Internally rotated or more han 10° externally rotated implants will be excluded. The rotation of femoral implant is measured on postoperative CT images in reference to surgical epicondylar line. The rotation of tibial implant is determined according to Berger's measurement)
12. Limb surgery within 3 months before the analysis
13. Postoperative revision surgery due to deep wound infection

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Knee Kinematics measured though all Degrees of freedom (DOF) | 1 year
  Roentgen Fluoroscopic Stereophotogrammetric Analysis (RFSA). We measure all DOFs (i.e. X-Y-Z rotations and translations in degrees and millimeters respectively)

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 1 year
  Patient Reported Outcome Measure (PROM)
Knee injury and Osteoarthritis Outcome Score (KOOS) | 1 year
  PROM
Forgotten Joint Score 12 (FJS-12) | 1 year
  PROM
Range of motion (ROM) | 1 year
  Clinical measurement using goniometer
Hip-knee-ankle angle (HKA-angle) | 1 year
  The axis of the lower extremity after knee arthroplasty
CT-rotation of implants | 1 year
  Evaluation of tibia implant rotation using Berger's method
Clinical stability | 1 year
  Varus-valgus stability in clinical testing

CONTACTS AND LOCATIONS:
Overall Officials: Frank-David Oehrn, MD, Principal Investigator — CIRRO and Kristiansund Hospital, Helse More and Romsdal Trust; Stephan Maximillian Røhrl, PhD, Study Director — CIRRO and Oslo University Hospital, Ullevål; Lars Harald William Engseth, MD, Principal Investigator — CIRRO and Oslo University Hospital, Ullevål
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Kurtz SM, Lau E, Ong K, Zhao K, Kelly M, Bozic KJ. Future young patient demand for primary and revision joint replacement: national projections from 2010 to 2030. Clin Orthop Relat Res. 2009 Oct;467(10):2606-12. doi: 10.1007/s11999-009-0834-6. Epub 2009 Apr 10. PMID 19360453
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Dieppe P, Lim K, Lohmander S. Who should have knee joint replacement surgery for osteoarthritis? Int J Rheum Dis. 2011 May;14(2):175-80. doi: 10.1111/j.1756-185X.2011.01611.x. PMID 21518317
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Wylde V, Jeffery A, Dieppe P, Gooberman-Hill R. The assessment of persistent pain after joint replacement. Osteoarthritis Cartilage. 2012 Feb;20(2):102-5. doi: 10.1016/j.joca.2011.11.011. Epub 2011 Nov 30. PMID 22178464
- [Background] Ravi B, Croxford R, Reichmann WM, Losina E, Katz JN, Hawker GA. The changing demographics of total joint arthroplasty recipients in the United States and Ontario from 2001 to 2007. Best Pract Res Clin Rheumatol. 2012 Oct;26(5):637-47. doi: 10.1016/j.berh.2012.07.014. PMID 23218428
- [Background] Ibrahim T, Bloch B, Esler CN, Abrams KR, Harper WM. Temporal trends in primary total hip and knee arthroplasty surgery: results from a UK regional joint register, 1991-2004. Ann R Coll Surg Engl. 2010 Apr;92(3):231-5. doi: 10.1308/003588410X12628812458572. Epub 2010 Mar 10. PMID 20223054
- [Background] Watanabe T, Ishizuki M, Muneta T, Banks SA. Knee kinematics in anterior cruciate ligament-substituting arthroplasty with or without the posterior cruciate ligament. J Arthroplasty. 2013 Apr;28(4):548-52. doi: 10.1016/j.arth.2012.06.030. Epub 2012 Oct 31. PMID 23122654
- [Background] Bell SW, Young P, Drury C, Smith J, Anthony I, Jones B, Blyth M, McLean A. Component rotational alignment in unexplained painful primary total knee arthroplasty. Knee. 2014 Jan;21(1):272-7. doi: 10.1016/j.knee.2012.09.011. Epub 2012 Nov 7. PMID 23140906
- [Background] Smith PN, Refshauge KM, Scarvell JM. Development of the concepts of knee kinematics. Arch Phys Med Rehabil. 2003 Dec;84(12):1895-902. doi: 10.1016/s0003-9993(03)00281-8. PMID 14669200
- [Background] Chalidis BE, Sachinis NP, Papadopoulos P, Petsatodis E, Christodoulou AG, Petsatodis G. Long-term results of posterior-cruciate-retaining Genesis I total knee arthroplasty. J Orthop Sci. 2011 Nov;16(6):726-31. doi: 10.1007/s00776-011-0152-1. Epub 2011 Sep 10. PMID 21909722
- [Background] Font-Rodriguez DE, Scuderi GR, Insall JN. Survivorship of cemented total knee arthroplasty. Clin Orthop Relat Res. 1997 Dec;(345):79-86. PMID 9418624
- [Background] Sabouret P, Lavoie F, Cloutier JM. Total knee replacement with retention of both cruciate ligaments: a 22-year follow-up study. Bone Joint J. 2013 Jul;95-B(7):917-22. doi: 10.1302/0301-620X.95B7.30904. PMID 23814243
- [Background] Price AJ, Waite JC, Svard U. Long-term clinical results of the medial Oxford unicompartmental knee arthroplasty. Clin Orthop Relat Res. 2005 Jun;(435):171-80. doi: 10.1097/00003086-200506000-00024. PMID 15930935
- [Background] Malchau H. Introducing new technology: a stepwise algorithm. Spine (Phila Pa 1976). 2000 Feb 1;25(3):285. doi: 10.1097/00007632-200002010-00004. No abstract available. PMID 10703097
- [Background] Malchau H, Bragdon CR, Muratoglu OK. The stepwise introduction of innovation into orthopedic surgery: the next level of dilemmas. J Arthroplasty. 2011 Sep;26(6):825-31. doi: 10.1016/j.arth.2010.08.007. Epub 2010 Oct 2. PMID 20888183
- [Background] Gao F, Henricson A, Nilsson KG. Cemented versus uncemented fixation of the femoral component of the NexGen CR total knee replacement in patients younger than 60 years: a prospective randomised controlled RSA study. Knee. 2009 Jun;16(3):200-6. doi: 10.1016/j.knee.2008.11.009. Epub 2008 Dec 19. PMID 19097910
- [Background] Iwaki H, Pinskerova V, Freeman MA. Tibiofemoral movement 1: the shapes and relative movements of the femur and tibia in the unloaded cadaver knee. J Bone Joint Surg Br. 2000 Nov;82(8):1189-95. doi: 10.1302/0301-620x.82b8.10717. PMID 11132285
- [Background] Pinskerova V, Johal P, Nakagawa S, Sosna A, Williams A, Gedroyc W, Freeman MA. Does the femur roll-back with flexion? J Bone Joint Surg Br. 2004 Aug;86(6):925-31. doi: 10.1302/0301-620x.86b6.14589. PMID 15330038
- [Background] Pinskerova V, Samuelson KM, Stammers J, Maruthainar K, Sosna A, Freeman MA. The knee in full flexion: an anatomical study. J Bone Joint Surg Br. 2009 Jun;91(6):830-4. doi: 10.1302/0301-620X.91B6.22319. PMID 19483242
- [Background] Nakagawa S, Kadoya Y, Todo S, Kobayashi A, Sakamoto H, Freeman MA, Yamano Y. Tibiofemoral movement 3: full flexion in the living knee studied by MRI. J Bone Joint Surg Br. 2000 Nov;82(8):1199-200. doi: 10.1302/0301-620x.82b8.10718. PMID 11132287
- [Background] Freeman MA, Pinskerova V. The movement of the knee studied by magnetic resonance imaging. Clin Orthop Relat Res. 2003 May;(410):35-43. doi: 10.1097/01.blo.0000063598.67412.0d. PMID 12771815
- [Background] Freeman MA, Pinskerova V. The movement of the normal tibio-femoral joint. J Biomech. 2005 Feb;38(2):197-208. doi: 10.1016/j.jbiomech.2004.02.006. PMID 15598446
- [Background] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091
- [Background] van Ijsseldijk EA, Lebel B, Stoel BC, Valstar ER, Gouzy S, Vielpeau C, Kaptein BL. Validation of the in vivo volumetric wear measurement for total knee prostheses in model-based RSA. J Biomech. 2013 Apr 26;46(7):1387-91. doi: 10.1016/j.jbiomech.2013.02.021. Epub 2013 Mar 26. PMID 23540721